CLINICAL TRIAL: NCT03580330
Title: Could Low-Cost Mobile Health Interventions Make a Difference?:Enhancing Outcomes of Noncommunicable Diseases Care in Rural Settings and Refugee Camps
Brief Title: Use of Low-cost mHealth Intervention to Enhance Outcomes of Noncommunicable Diseases Care in Rural and Refugee Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: International Development Research Centre, Canada (Other Government); Ministry of Public Health (MOPH), Lebanon (Unknown); United Nations Relief and Works Agency (UNRWA) (Unknown)
Responsible Party: Principal Investigator, Shadi Saleh, Director, Global Health Institute, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: FHS.SS.11
Record Dates: First submitted 2018-06-01; First posted 2018-07-09 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: noncommunicable diseases; hypertension; diabetes mellitus; telemedicine; mobile health; rural health; refugees
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: This study reports on a community trial in which PHC centers, along their respective catchment areas, were randomly allocated into control and intervention sites with the aim of assessing the change in selected NCD care quality indicators (QIs) among community individuals and patients. Patients in the intervention sites received a 1-year mHealth intervention, and their pre- and postintervention outcomes were assessed through measurement of QIs. Patients in the control sites received no intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: mHealth intervention
- Control Group (No Intervention)

INTERVENTIONS:
Other: mHealth intervention — Individual in the intervention group receive a weekly educational health SMS for the intervention period of 1 year. SMS content covered different health themes providing health information on lifestyle, dietary habits, body weight, smoking, medications, importance of compliance, as well as symptoms and self-management of HTN and diabetes. Community individuals who were diagnosed and were receiving necessary care previous to the investigator's intervention were sent weekly informative health SMS, as well as customized SMSs reminders to follow up on their scheduled medical appointments (eg, to check their HbA1c levels and have their annual foot or eye exams).
  Arms: Intervention Group

SUMMARY:
Rural areas and refugee camps are characterized by poor access of patients to needed noncommunicable disease (NCD)-related health services, including diabetes and hypertension. This community trial study aims to assess the effect of employing low-cost mHealth tools on the accessibility to health services and improvement of health indicators of individuals with NCDs in rural areas and refugee camps in Lebanon.

DETAILED DESCRIPTION:
Rural areas and refugee camps are characterized by poor access of patients to needed noncommunicable disease (NCD)-related health services, including diabetes and hypertension. Employing low-cost innovative eHealth interventions, such as mobile health (mHealth), may help improve NCDs prevention and control among disadvantaged populations.

The aim of this study was to assess the effect of employing low-cost mHealth tools on the accessibility to health services and improvement of health indicators of individuals with NCDs in rural areas and refugee camps in Lebanon.

This is a community trial study in which centers were allocated randomly into control and intervention sites. The effect of an employed mHealth intervention is assessed through selected quality indicators examined in both control and intervention groups. Sixteen primary health care centers (eight controls, eight interventions) located in rural areas and Palestinian refugee camps across Lebanon were included in this study. Data on diabetic and hypertensive patients-1433 in the intervention group and 926 in the control group-was extracted from patient files in the pre and postintervention periods. The intervention entailed weekly short message service messages, including medical information, importance of compliance, and reminders of appointments or regular physician follow-up. Internationally established care indicators were utilized in this study.

ELIGIBILITY:
Inclusion Criteria:

* Registered at the Primary Healthcare Center as diabetics and/or hypertensive or diagnosed with or suspected to have diabetes and/or hypertension
* Aged 40 years or more
* Lebanese or Palestinian nationality

Exclusion Criteria:

* aged less than 40 years
* Non-Lebanese / Non-Palestinian
* No exclusion based on gender, educational and literacy level, disability, or presence of other medical conditions

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2359 (Actual)
Dates: Start 2014-04-17 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Control (blood pressure (SBP/DBP) <140/90 mmHg)) | At 1 year from the time of initiation of the intervention
  blood pressure (SBP/DBP) <140/90 mmHg
Mean HbA1c | At 1 year from the time of initiation of the intervention
  HbA1c level assessed for each patient

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Saleh S, Farah A, Dimassi H, El Arnaout N, Constantin J, Osman M, El Morr C, Alameddine M. Using Mobile Health to Enhance Outcomes of Noncommunicable Diseases Care in Rural Settings and Refugee Camps: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jul 13;6(7):e137. doi: 10.2196/mhealth.8146. PMID 30006326